CLINICAL TRIAL: NCT02091349
Title: Tolerance and Utilization of Polydextrose, Inulin, and Soluble Corn Fiber
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Urbana-Champaign (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 09491
Record Dates: First submitted 2014-03-17; First posted 2014-03-19 (Estimated); Last update posted 2014-05-14 (Estimated); Status verified 2014-05

CONDITIONS: Tolerance
MeSH Terms: interventions — polydextrose

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group A- placebo (Placebo Comparator): control- snack bar or muffin containing no fiber
  Interventions: Other: polydextrose; Other: soluble corn fiber
- Group B- polydextrose (Experimental): polydextrose- randomly bonded polysaccharide of glucose which is poorly digested in small intestine
  Interventions: Other: polydextrose; Other: soluble corn fiber
- Group C- soluble corn fiber (Experimental): Soluble corn fiber made from corn starch and contains oligosaccharides with random glyucosyl bonds and may contain minor amounts of monosaccharides
  Interventions: Other: polydextrose; Other: soluble corn fiber

INTERVENTIONS:
Other: polydextrose — polydextrose- 7, 14, or 21 grams/day 3X3 latin square with 3 periods
Other: soluble corn fiber — nutirose- 7, 14, or 21 grams/day

SUMMARY:
The objective of this study is to determine the tolerance and utilization of polydextrose and soluble corn fiber through analyses of fecal samples of fermentative end-products (short-chain fatty acids, ammonia, phenol, and indole) and shifts in microbial populations.

DETAILED DESCRIPTION:
Soluble fibers have been shown to have many positive effects in humans, including laxation and maintaining gastrointestinal health. It is expected that feeding soluble fibers will decrease protein fermentative end=products while increasing carbohydrate fermenative end-products, and lead to a more beneficial microbial profile. Determination of the effects of nutriose and polydextrose when included as supplemental fiber in a human diet will give insights to its potential to maintain or improve gut health and highlight its use in the food industry.

The object of this study are first to determine the tolerance of soluble fibers polydextrose, inulin and nutriose when provided as supplemental fiber to an existing diet. The second objective is to determine the utilization of polydextrose and nutriose through analyses of fecal samples of fermentative end-products and shifts in microbial populations.

ELIGIBILITY:
Inclusion Criteria:

* have body mass index (BMI) between 18.5 and 31 kg/m2
* free of metabolic and gastrointestinal disease

Exclusion Criteria:

* BMI less than 18.5 or greater than 31 kg/m2
* presence of metabolic or gastrointestinal diseases

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2010-07; Primary Completion 2011-01 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
Fecal bacteria | Days 16-21 of each treatment period
  Fecal samples will be collected on days 16-21 of each treatment period. Participants were provided fecal collection materials (fecal hats, packs, and Ziploc bags). Within 15 minutes of defecation, participants will bring their fecal sample to the designated collection site then be processed by a team. Fecal specimens will be aliquoted into containers for analysis of bacterial species present.
Fecal fermentation end products | Days 16-21 of each treatment period
  Fecal samples will be collected on days 16-21 of each treatment period. Participants were provided fecal collection materials (fecal hats, packs, and Ziploc bags). Within 15 minutes of defecation, participants will bring their fecal sample to the designated collection site then be processed by a team. Fecal specimens will be aliquoted into containers for fermentation end product analysis (short-chain fatty indoles, ammonia) and dry matter.

SECONDARY OUTCOMES:
Gastrointestinal Tolerance | Daily during each 21 day treatment period
  Gastrointestinal tolerance was scored using the following scale: 1=absent, 2=mild, 3=moderate, 4=severe. All study participants booklets with daily tolerance questionnaires in them. The participants will complete the questionnaires on their own each day.
Daily Stool Characteristics | Daily during each 21 day treatment period
  Participants are provided a journal to complete on their own each day, a questionnaire about their stool characteristics. Participants were score the ease of stool passage using the following scale: 1=very easy, 2=easy, 3=neither easy nor difficult, 4=difficult, 5=very difficult.
  Stool consistency was scored using the Bristol stool scale: 1=separate hard lumps, like nuts; 2=sausage-shaped but lumpy; 3=like a sausage cracks on surface; 4=Like a sausage or snake, smooth and soft; 5=soft blobs with clear-cut edges; 6=fluffy pieces with ragged edges, 7=watery, no solid pieces, entirely liquid.

OTHER OUTCOMES:
Daily food intake journals | Daily during each 21-day treatment period
  Participants were provided a journal to record their daily food and beverage intake. Each week the participants met with a study personnel minutes to review the journal and turn it in.

CONTACTS AND LOCATIONS:
Overall Officials: George Fahey, Jr, PhD, Principal Investigator — UIUC

REFERENCES:
- [Derived] Holscher HD, Caporaso JG, Hooda S, Brulc JM, Fahey GC Jr, Swanson KS. Fiber supplementation influences phylogenetic structure and functional capacity of the human intestinal microbiome: follow-up of a randomized controlled trial. Am J Clin Nutr. 2015 Jan;101(1):55-64. doi: 10.3945/ajcn.114.092064. Epub 2014 Nov 12. PMID 25527750